CLINICAL TRIAL: NCT06591273
Title: Efficacy and Safety of Infliximab Biosimilar in Treatment of Moderate to Severe Psoriasis; A Single-arm Clinical Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Hira Tariq, Dr, Services Institute of Medical Sciences, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2023/1201/SIMS
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
Keywords: Infliximab biosimilar, Remsima, Plaque psoriasis, Biologics
MeSH Terms: interventions — CT-P13

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult Patients of moderate to severe plaque psoriasis (Experimental)
  Interventions: Biological: Infliximab-dyyb Biosimilar (Remsima)

INTERVENTIONS:
Biological: Infliximab-dyyb Biosimilar (Remsima) — Subcutaneous injections of Infliximab-dyyb Biosimilar (Remsima) were injected weekly for 4 weeks and then fortnightly for 24 weeks

SUMMARY:
The goal of this clinical trial is to learn if Infliximab Biosimilar Remsima works to treat moderate to severe plaque Psoriasis in adults. It will also learn about the safety of the drug. The main questions it aims to answer are:

Does Infliximab-dyyb Biosimilar (Remsima) works to treat moderate to severe plaque Psoriasis in adults in reducing disease severity and relapses? What medical problems do participants have when taking Remsima?

Participants will:

be injected Infliximab Biosimilar Remsima weekly for 4 weeks and then fortnightly till 24 weeks They will be followed for efficacy and safety and lab tests at week 4, 14, 24 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients of moderate to severe plaque psoriasis Biologically naive patients

Exclusion Criteria:

* Patients with active or latent TB, Hepatitis B or C, HIV. Immunocompromised patients due to drugs or disease. Patients on systemic anti-psoriastic medications in last three months. Patients with personal or strong family history of heart disease. Any other medical comorbidity (hepatic or renal) or contraindication to biologic/ biosimilars.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
At least 50% reduction in PASI | 14 weeks
  PASI should reduce to at least 50% of baseline (pre-treatment)
At least 50% reduction in DLQI | 14 weeks
  DLQI (Dermatology Life Quality Index) should reduce to at least 50% of baseline (pre-treatment)

SECONDARY OUTCOMES:
Maintenance of At least 50% reduction in PASI and DLQI | 24 weeks
  Maintenance of At least 50% reduction in PASI and DLQI from baseline (pre-treatment)
Maintenance of At least 50% reduction in PASI and DLQI | 52 weeks
  Maintenance of At least 50% reduction in PASI and DLQI from baseline (pre-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hira Tariq, MBBS, FCPS Derma, Principal Investigator — Services Institute of Medical Sciences, Pakistan
Locations (1):
- Department of Dermatology, Services Institute of Medical Sciences/ Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6661374/